CLINICAL TRIAL: NCT03636971
Title: Gait Analysis Following Single-shot Hyaluronic Acid Supplementation: a Pilot Randomised Double-blinded Clinical Trial
Brief Title: Gait Analysis Following Knee Viscosupplementation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigitte Jolles, MD (Other)
Responsible Party: Sponsor-Investigator, Brigitte Jolles, MD, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: CER-VD No 273/13
Record Dates: First submitted 2018-08-06; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Gait; Knee Osteoarthritis; Injection
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid; Mannitol; Sorbitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hyaluronic acid with mannitol (Experimental)
  Interventions: Drug: hyaluronic acid with mannitol
- hyaluronic acid with sorbitol (Experimental)
  Interventions: Drug: hyaluronic acid with sorbitol
- saline (Active Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: hyaluronic acid with mannitol — single shot injection (Ostenil Plus®, TRB Chemedica SA, CH, 1800kD)
  Arms: hyaluronic acid with mannitol
Drug: hyaluronic acid with sorbitol — single shot injection (Synolis®, Gebro-Pharma AG, CH, 2000 kD)
  Arms: hyaluronic acid with sorbitol
Drug: Placebos — single shot injection of saline, same volume
  Arms: saline

SUMMARY:
This is a pilot, double-blind, randomised trial that investigates which gait parameters are more sensitive following a single bolus injection of hyaluronic acid with mannitol, hyaluronic acid with sorbitol, or saline placebo for knee osteoarthritis. Outcome measures are gait analysis through a inertial sensors (Physilog), Knee Society Score (KSS), University of California Los Angeles (UCLA) activity-scale and EuroQol 5Dimensions. Follow-up will be of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary knee OA Ahlbäck II-III and signed consent forms.

Exclusion Criteria:

* recent history of infection, diabetes, neurological impairment, chronic venous or lymphatic stasis, pain medication of level 2 or 3, psychiatric conditions, contraindications for HA joint injection and previous HA or steroid injections in the last six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Gait Speed | 4 weeks following injection
  measured over the 30m of the test trial using an inertial-based system (Physilog, BioAGM, CH) following a previously validated protocol. Spatiotemporal parameters are analysed (i.e. gait speed, cadence, limping...)

SECONDARY OUTCOMES:
KSS specific knee mobility scale | 4 weeks following injection
  Knee specific clinician-based mobility scale based on clinical examination. Score interpretation: 80-100 Excellent, Score 70-79 Good, Score 60-69 Fair, score below 60 Poor.
EuroQool -5 dimensions self-reported scale of quality of life | 4 weeks following injection
  The EQ-5D-5L essentially consists on the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises 5dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.Each dimension comprising the EQ-5D descriptive system is divided into 5levels of perceived problems:Level 1:no problem Level 2:slight problems Level 3: moderate problems Level 4:severe problems Level 5: extreme problems. A unique health state is defined by combining 1 level from each of the 5 dimensions.A total of 3125 possible health states is defined in this way. Each state is referred to in terms of a 5 digit code.
  The EQ VAS records the patient's self-rated health on a 20cm vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
UCLA- activity scale | 4 weeks following injection
  Activity numerical ordinal scale ranging from 1 (lowest) to 10 (highest)
Visual Analogue Scale (VAS) pain | 4 weeks following injection
  continual numerical scale (0-10), 0 the best score (no pain) and 10 the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Brigitte, Study Chair — CHUV
Locations (1):
- CHUV - Hopital Orthopedique, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pereira LC, Schweizer C, Moufarrij S, Krahenbuhl SM, Favre J, Gremion G, Applegate LA, Jolles BM. Gait analysis following single-shot hyaluronic acid supplementation: a pilot randomized double-blinded controlled trial. Pilot Feasibility Stud. 2019 Apr 22;5:56. doi: 10.1186/s40814-019-0443-4. eCollection 2019. PMID 31024734